CLINICAL TRIAL: NCT06314646
Title: Postoperative and Long-term Outcomes of Transanal Tran-section and Single-stapled Anastomosis (TTSS) in Rectal Can-cer Patients: a Multicentric International IDEAL Stage 2b Prospective Parallel Cohort Study
Brief Title: Transanal Transection and Single-stapled Anastomosis (TTSS) in Rectal Cancer Patients
Acronym: TTSS-REC
Status: Recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 3747
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Rectal Cancer; Surgery
Keywords: Rectal Cancer; Transanal Transection and Single-Stapled anastomosis; Total Mesorectal Excision
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transanal Transection and Single-Stapled anastomosis (TTSS): Patients will undergo rectal cancer surgery through low rectal resection with Transanal Transection and Single-Stapled anastomosis (TTSS)
  Interventions: Procedure: Transanal Transection and Single-Stapled anastomosis (TTSS)
- Double-stapled Total Mesorectal Excision (TME): Patients will undergo rectal cancer surgery through low rectal resection with double-stapled anastomosis Total Mesorectal Excision (TME)
  Interventions: Procedure: Double-stapled Total Mesorectal Excision (TME)

INTERVENTIONS:
Procedure: Transanal Transection and Single-Stapled anastomosis (TTSS) — Low anterior rectal resection with Transanal Transection and Single-Stapled anastomosis (TTSS)
  Groups: Transanal Transection and Single-Stapled anastomosis (TTSS)
Procedure: Double-stapled Total Mesorectal Excision (TME) — Low anterior rectal resection with double-stapled Total Mesorectal Excision (TME)
  Groups: Double-stapled Total Mesorectal Excision (TME)

SUMMARY:
The Transanal Transection and Single-Stapled anastomosis (TTSS) technique may be a valid alternative to traditional double-stapled anastomosis for low rectal cancer surgery. This study aims to compare the postoperative and functional outcomes of patients receiving TTSS and traditional double-stapled anastomosis.

DETAILED DESCRIPTION:
The Transanal Transection and Single-Stapled anastomosis (TTSS) technique has become a valid alternative to the standard double-stapled anastomosis approach in the surgical treatment of low rectal cancer. Recent evidence showed a significantly reduced number of anastomotic leaks in patients undergoing TTSS compared with patients receiving double-stapled anastomosis, suggesting that TTSS may be technically feasible and may provide a surgical advantage over the traditional double-stapled technique. However, these studies were severely limited by their single-center and retrospective nature. This study aims to confirm the retrospective findings by extending the data collection to additional countries and provide prospective data collection.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years old) patients, men and women, diagnosed with rectal cancer scheduled for elective rectal resection with Total Mesorectal Excision (TME) with double-stapled or Transanal Transection and Single-Stapled anastomosis (TTSS) approaches.
* Patients scheduled for open, laparoscopic, or robotic surgery.
* Patients preoperatively indicated for sphincter-saving procedures with or without protective-stoma.

Exclusion Criteria:

* Immediate or delayed hand-sewn coloanal anastomosis.
* Patients requiring abdominoperineal resection (APR). Patients undergoing unplanned non-reconstructive surgery will be withdrawn from the study.
* Patients with concurrent or previous invasive pelvic malignant tumors. Patients with an intraoperative evidence of invasive pelvic malignant tumors will be withdrawn from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients diagnosed with rectal cancer scheduled for elective rectal resection with double-stapled or Transanal Transection and Single-Stapled anastomosis (TTSS).
Sampling Method: Non-Probability Sample
Enrollment: 472 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of anastomotic leak | 90 days after surgery
  Rate difference of clinical and/or radiological anastomotic leaks in the study cohorts.

SECONDARY OUTCOMES:
Rate of postoperative complications | 90 days after surgery
  Rate difference of overall postoperative complications- classified according to the Clavien-Dindo scale [ranging from 0 (no complications) to 5 (complications leading to death)]- in the study cohorts.
Postoperative Recovery Profile (PRP) score | 90 days after surgery
  Median difference of Postoperative Recovery Profile (PRP) [ranging from 0 (completely recovered) to 68 (not recovered)] in the study cohorts.
Proportion of patients fit for stoma closure | 12 months after surgery
  Proportion difference of patients fit for stoma closure in the study cohorts. Patients fit for stoma closure have already closed the stoma or have an intact anastomosis as demonstrated by a water contrast enema, Computed Tomography (CT) scan, endoscopic, or surgical revision.
Healthcare costs | 12 months after surgery
  Median difference of healthcare costs (direct and indirect) in the study cohorts.
Low Anterior Resection Syndrome (LARS) score | 6 months after surgery or stoma closure
  Median difference of Low Anterior Resection Syndrome (LARS) score [ranging from 0 (no LARS symptoms) to 42 (severe LARS symptoms)] in the study cohorts.
Low Anterior Resection Syndrome (LARS) score | 12 months after surgery or stoma closure
  Median difference of Low Anterior Resection Syndrome (LARS) score [ranging from 0 (no LARS symptoms) to 42 (severe LARS symptoms)] in the study cohorts.
Low Anterior Resection Syndrome (LARS) score | 24 months after surgery or stoma closure
  Median difference of Low Anterior Resection Syndrome (LARS) score [ranging from 0 (no LARS symptoms) to 42 (severe LARS symptoms)] in the study cohorts.
Cancer recurrence | 24 months after surgery
  Incidence rate difference of cancer recurrence- defined as any local or distal recurrence or metastasis- in the study cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Spinelli, MD, PhD, Principal Investigator — IRCCS Huamanitas Research Hospital
Locations (1):
- IRCCS Humanitas Research Hospital, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No